CLINICAL TRIAL: NCT03122860
Title: A Phase 2, 24-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of SM04690 for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Brief Title: A Study Evaluating the Safety and Efficacy of SM04690 for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04690-OA-04
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Samumed
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 0.03 mg SM04690 (Experimental): Single intra-articular injection of 0.03 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690
- 0.07 mg SM04690 (Experimental): Single intra-articular injection of 0.07 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690
- 0.15 mg SM04690 (Experimental): Single intra-articular injection of 0.15 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690
- 0.23 mg SM04690 (Experimental): Single intra-articular injection of 0.23 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690
- Placebo (Placebo Comparator): Single intra-articular injection of 0 mg SM04690 in 2 mL vehicle
  Interventions: Other: Placebo
- Sham (Sham Comparator): Single intra-articular injection of 0 mg SM04690 in 0 mL vehicle
  Interventions: Other: Sham

INTERVENTIONS:
Drug: SM04690 — Healthcare professional-administered intra-articular injection performed once on Day 1 of the study
  Arms: 0.03 mg SM04690; 0.07 mg SM04690; 0.15 mg SM04690; 0.23 mg SM04690
Other: Placebo — Healthcare professional-administered intra-articular injection performed once on Day 1 of the study
  Arms: Placebo
Other: Sham — Healthcare professional-administered intra-articular injection performed once on Day 1 of the study
  Arms: Sham

SUMMARY:
This phase 2 study is a placebo-controlled, double-blind, parallel group study of four concentrations of SM04690 (0.03, 0.07, 0.15, and 0.23 mg per 2 mL injection) injected intraarticularly (IA) into the target knee joint of subjects with moderately to severely symptomatic osteoarthritis (OA). Based on previous studies of SM04690, key phenotypes of laterality (unilateral vs bilateral) as well as chronic pain (as measured by the Widespread Pain Index) were identified as confounding variables impacting the overall assessment of both radiologic and clinical efficacy outcomes. The design of SM04690-OA-04 is based upon previous study designs while assessing strategies to combat the confounding impact of laterality and chronic pain. To evaluate the effect of IA vehicle injection on patient-reported outcomes (PRO) such as pain, stiffness, and function in OA, this study also includes one cohort that receives a 2 mL IA injection of vehicle (placebo), and one cohort that receives a sham injection (i.e., a needle stick with 0 mL vehicle injected).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at screening (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
* Pain compatible with OA of the knee(s) for at least 26 weeks prior to screening
* Primary source of pain throughout the body is due to OA in the target knee
* Willingness to use an electronic diary on a daily basis in the evening for the screening period and 24-week study duration
* Negative drug test for opioids and drugs of abuse, except alcohol and marijuana, at screening
* Subjects with depression or anxiety must be clinically stable for 12 weeks prior to screening, and, if on treatment for depression or anxiety, be on 12 weeks of stable therapy
* Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
* Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed

Exclusion Criteria:

* Women who are pregnant, lactating, or have a positive pregnancy result at screening
* Women of child bearing potential who are sexually active and are not willing to use a highly effective method of birth control during the study period
* Males who are sexually active and have a partner who is capable of becoming pregnant, neither of whom have had surgery to become sterilized or whom are not using a highly effective method of birth control
* Body mass index (BMI) > 35
* Partial or complete joint replacement in either knee
* Currently requires regular use of ambulatory assistive devices (e.g., wheelchair, parallel bars, walker, canes, or crutches) or use of a lower extremity prosthesis, and/or a structural knee brace
* Previous participation in a Samumed clinical trial investigating SM04690
* Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to screening
* Any planned surgery during the study period
* History of malignancy within the last 5 years; however, subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible if completely excised. Subjects with other malignancies are eligible if they have been continuously disease free for at least 5 years prior to any study injection
* Comorbid conditions that could affect study endpoint assessments of the target knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout or pseudogout, and fibromyalgia
* Any diagnosed psychiatric condition that includes, but is not limited to, a history of mania, bipolar disorder, psychotic disorder, schizophrenia, schizoaffective disorder, major depressive disorder, or generalized anxiety disorder
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure, or an observational research trial related to osteoarthritis within 8 weeks prior to any study injection, or planned participation in any such trial
* Treatment of the target knee with intra-articular glucocorticoids (e.g., methylprednisolone) within 12 weeks prior to screening
* Any intra-articular injection into the target knee with a therapeutic aim including, but not limited to, viscosupplementation (e.g., hyaluronic acid), platelet-rich plasma (PRP), and stem cell therapies within 24 weeks prior to screening; treatment of the target knee with intra-articular glucocorticoids greater than 12 weeks prior to screening is allowed
* Treatment with systemic glucocorticoids greater than 10 mg prednisone or the equivalent per day within 4 weeks prior to screening
* Effusion of the target knee clinically requiring aspiration within 12 weeks prior to screening
* Use of electrotherapy, acupuncture, and/or chiropractic treatments for knee OA within 4 weeks prior to screening
* Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of intra-articular infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at study start
* Use of centrally acting analgesics (e.g., duloxetine) within 12 weeks prior to screening
* Use of anticonvulsants within 12 weeks prior to screening, unless used for seizure or migraine prophylaxis
* Subjects requiring the usage of opioids >1x per week within 12 weeks prior to screening
* Use of topical local anesthetic agents (gels, creams, or patches such as the Lidoderm patch) for the treatment of knee OA within 7 days of screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (71):
- United States (71):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Canoga Park, California
  - Research Site, Carmichael, California
  - Research Site, Cerritos, California
  - Research Site, El Cajon, California
  - Research Site, Gold River, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Rancho Mirage, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Marcos, California
  - Research Site, Spring Valley, California
  - Research Site, Boulder, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, DeLand, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Newton, Kansas
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Jefferson, Louisiana
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Troy, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, State College, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Angelo, Texas
  - Research Site, Arlington, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yazici Y, McAlindon TE, Gibofsky A, Lane NE, Lattermann C, Skrepnik N, Swearingen CJ, Simsek I, Ghandehari H, DiFrancesco A, Gibbs J, Tambiah JRS, Hochberg MC. A Phase 2b randomized trial of lorecivivint, a novel intra-articular CLK2/DYRK1A inhibitor and Wnt pathway modulator for knee osteoarthritis. Osteoarthritis Cartilage. 2021 May;29(5):654-666. doi: 10.1016/j.joca.2021.02.004. Epub 2021 Feb 12. PMID 33588087
- [Derived] Tambiah J, Kennedy S, Swearingen C, McAlindon T, Yazici Y. Impact of structural severity on outcomes in knee osteoarthritis: an analysis of data from phase 2 and phase 3 lorecivivint clinical trials. Rheumatology (Oxford). 2025 May 1;64(5):2583-2590. doi: 10.1093/rheumatology/keae610. PMID 39495154
- [Derived] Tambiah JRS, Simsek I, Swearingen CJ, Kennedy S, Cole BJ, McAlindon TE, Yazici Y. Comparing Patient-Reported Outcomes From Sham and Saline-Based Placebo Injections for Knee Osteoarthritis: Data From a Randomized Clinical Trial of Lorecivivint. Am J Sports Med. 2022 Mar;50(3):630-636. doi: 10.1177/03635465211067201. Epub 2022 Jan 10. PMID 35005990
- [Derived] Tambiah JRS, Kennedy S, Swearingen CJ, Simsek I, Yazici Y, Farr J, Conaghan PG. Individual Participant Symptom Responses to Intra-Articular Lorecivivint in Knee Osteoarthritis: Post Hoc Analysis of a Phase 2B Trial. Rheumatol Ther. 2021 Jun;8(2):973-985. doi: 10.1007/s40744-021-00316-w. Epub 2021 Jun 8. PMID 34101138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set (FAS) includes all subjects who were randomized and received a study injection, analyzed as randomized.
Pre-assignment Details: The Safety Analysis Set (SAS) [see 'Adverse Events' section] includes all subjects who received a study injection, analyzed as treated. Discrepancy in subject counts between FAS and SAS is the result of subjects who received a treatment that is different from the planned treatment group as randomized. Subjects who received a study treatment not as prescribed in the pharmacy manual are summarized in the "Other" treatment group for safety analysis reporting.
Period: Overall Study
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Started | 117 | 116 | 117 | 116 | 117 | 117
Full Analysis Set | 116 | 115 | 115 | 116 | 116 | 117
Completed | 107 | 111 | 105 | 105 | 102 | 105
Not Completed | 10 | 5 | 12 | 11 | 15 | 12
Not completed — Discontinued Before Treatment | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 2 | 3 | 3 | 5 | 4
Not completed — Subject Non-Compliance | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 5 | 7 | 9 | 8

BASELINE CHARACTERISTICS:
Population: All subjects who were randomized and received a study injection, analyzed as randomized (Full Analysis Set [FAS]). FAS is used to describe the analysis set which is as complete as possible and as close as possible to the intent-to-treat ideal of including all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham | Total
Number analyzed (Participants) | 116 | 115 | 115 | 116 | 116 | 117 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.9) | 59.9 (8.6) | 58.4 (8.3) | 58.5 (9.0) | 60.1 (9.0) | 59.0 (8.0) | 59.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 66 | 69 | 61 | 64 | 70 | 406
  Male | 40 | 49 | 46 | 55 | 52 | 47 | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 22 | 10 | 16 | 24 | 115
  Not Hispanic or Latino | 95 | 93 | 93 | 106 | 100 | 93 | 580
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2 | 2 | 6
  Asian | 5 | 5 | 6 | 5 | 6 | 3 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 0 | 0 | 1 | 2 | 6
  Black or African American | 24 | 22 | 25 | 21 | 17 | 24 | 133
  White | 85 | 83 | 84 | 89 | 90 | 86 | 517
  More than one race | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Population: BMI was not collected for one participant in the 0.03 mg SM04690 cohort.
  kg/m²
    number analyzed (Participants) | 115 | 115 | 115 | 116 | 116 | 117 | 694
    (all) | 29.17 (3.76) | 29.14 (3.64) | 29.38 (4.10) | 28.53 (4.39) | 28.62 (4.29) | 28.97 (3.84) | 28.97 (4.01)
Kellgren-Lawrence Grade [Count of Participants; unit: Participants] — Participants' knee osteoarthritis was graded in accordance with the following definitions of Kellgren-Lawrence Grade: None (Grade 0) - Normal appearance of the knee; Doubtful (Grade 1): Doubtful narrowing of joint space and possible osteophytic lipping; Minimal (Grade 2): Definite osteophytes and possible narrowing of joint space; Moderate (Grade 3): Moderate multiple osteophytes, definite narrowing of the joint space, some sclerosis and possible deformity of bone ends; Severe (Grade 4): Large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.
  Participants
    Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Grade 2 | 53 | 38 | 47 | 53 | 43 | 57 | 291
    Grade 3 | 63 | 74 | 68 | 63 | 72 | 58 | 398
    Grade 4 | 0 | 2 | 0 | 0 | 1 | 2 | 5
Osteoarthritis Laterality [Count of Participants; unit: Participants]
  Unilateral | 59 | 62 | 63 | 63 | 61 | 62 | 370
  Bilateral | 57 | 53 | 52 | 53 | 55 | 55 | 325
Widespread Pain (WP) [Count of Participants; unit: Participants] — Subjects were required to complete the Widespread Pain Index & Symptom Severity questionnaire. The Widespread Pain Index (WPI) is a body map consisting of 19 prespecified areas where subjects can indicate the presence of pain during the past seven days with a possible score 0-19. Question 2 of the Symptom Severity section of the questionnaire (SSQ2) focuses on the presence and severity of three prespecified symptoms (fatigue, trouble thinking or remembering, and waking up tired) during the past seven days with a possible score of 0-9. WP+: WPI > 4 and/or SSQ2 > 2, WP-: WPI <= 4 and SSQ2 <= 2
  Participants
    WP- | 92 | 93 | 90 | 93 | 93 | 94 | 555
    WP+ | 24 | 22 | 25 | 23 | 23 | 23 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Osteoarthritis (OA) Pain in the Target Knee as Assessed by the Weekly Average of Daily Pain Numeric Rating Scale (NRS)
Description: Change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 24. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain (pain as bad as one can imagine).
Time Frame: Baseline and Week 24
Population: Data is reported as observed with no imputation. Discrepancy between the number of participants analyzed and the number of participants assigned to the arms is the result of missing data and/or subject withdrawal.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 98 | 102 | 92 | 90 | 95 | 91
score on a scale | -2.77 (2.44) | -2.93 (2.21) | -2.43 (2.18) | -3.03 (2.43) | -2.26 (2.44) | -2.21 (2.46)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.179, ANCOVA; Median Difference (Final Values) = -0.46, 95% CI 2-sided [-1.13 to 0.21]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.031, ANCOVA; Median Difference (Final Values) = -0.70, 95% CI 2-sided [-1.34 to -0.06]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.675, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.81 to 0.52]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.022, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.51 to -0.12]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.780, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.79 to 0.59]

2. Primary Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscore (WOMAC Pain)
Description: Change from baseline OA pain in the target knee as assessed by WOMAC Numeric Rating Scale (NRS 3.1) pain subscore (WOMAC Pain) at Week 24. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore is standardized and reported ranging from 0 to 100 [0 = no pain; 100 = pain as bad as it can be].
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 94 | 102 | 93 | 93 | 93 | 92
score on a scale | -27.6 (22.8) | -30.0 (22.5) | -24.7 (21.6) | -33.3 (22.9) | -25.5 (25.8) | -22.5 (24.6)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.612, ANCOVA; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-8.32 to 4.91]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.223, ANCOVA; Mean Difference (Final Values) = -4.01, 95% CI 2-sided [-10.47 to 2.46]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.590, ANCOVA; Mean Difference (Final Values) = 1.84, 95% CI 2-sided [-4.89 to 8.57]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.031, ANCOVA; Mean Difference (Final Values) = -7.36, 95% CI 2-sided [-14.03 to -0.69]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.403, ANCOVA; Mean Difference (Final Values) = -2.89, 95% CI 2-sided [-9.70 to 3.92]

3. Primary Outcome: Change From Baseline OA Function in the Target Knee as Assessed by WOMAC Physical Function Subscore (WOMAC Function)
Description: Change from baseline OA function in the target knee as assessed by WOMAC Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function) at Week 24. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore is standardized and reported ranging from 0 to 100 [0 = no functional disability, 100 = unable to function].
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 94 | 102 | 93 | 93 | 93 | 92
score on a scale | -27.7 (21.1) | -29.3 (23.0) | -23.6 (21.6) | -32.4 (22.1) | -24.9 (23.7) | -23.8 (23.7)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.432, ANCOVA; Mean Difference (Final Values) = -2.58, 95% CI 2-sided [-9.04 to 3.88]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.180, ANCOVA; Mean Difference (Final Values) = -4.34, 95% CI 2-sided [-10.69 to 2.02]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.718, ANCOVA; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-5.33 to 7.72]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.017, ANCOVA; Mean Difference (Final Values) = -7.99, 95% CI 2-sided [-14.54 to -1.45]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.682, ANCOVA; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-8.06 to 5.29]

4. Primary Outcome: Change From Baseline in Medial Joint Space Width (mJSW) of the Target Knee
Description: Change from baseline in mJSW as documented by radiograph of the target knee.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 104 | 109 | 103 | 101 | 96 | 104
mm | 0.02 (0.72) | -0.11 (0.53) | -0.11 (0.92) | -0.03 (0.45) | -0.01 (0.60) | -0.08 (0.58)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.822, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.16 to 0.21]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.162, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.27 to 0.04]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.267, ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.34 to 0.09]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.685, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.18 to 0.12]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.342, ANCOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.09 to 0.24]

5. Secondary Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment (PtGA)
Description: Change from baseline OA disease activity as assessed by PtGA at Week 24. The PtGA was completed using a 100 mm visual analog scale (VAS) adapted from the Patient Assessment Form © 1999, American College of Rheumatology. The subject rated how well he/she was doing, considering all the ways in which illness and health conditions may affected him/her. The VAS scale was anchored by "Very Well" on the left (scored as 0) and "Very Poorly" on the right (scored as 100). Higher scores indicated poorer disease assessment by the subject.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 90 | 99 | 92 | 92 | 90 | 90
mm | -16.0 (23.5) | -19.8 (27.1) | -11.9 (27.5) | -18.3 (24.5) | -13.0 (21.6) | -13.8 (24.4)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.500, ANCOVA; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-8.36 to 4.10]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.082, ANCOVA; Mean Difference (Final Values) = -5.54, 95% CI 2-sided [-11.80 to 0.72]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.552, ANCOVA; Mean Difference (Final Values) = -1.94, 95% CI 2-sided [-8.36 to 4.48]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.033, ANCOVA; Mean Difference (Final Values) = -6.86, 95% CI 2-sided [-13.16 to -0.56]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.887, ANCOVA; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-5.79 to 6.68]

6. Other Pre Specified Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by WOMAC Pain Subscore (WOMAC Pain)
Description: Change from baseline OA pain in the target knee as assessed by WOMAC Numeric Rating Scale (NRS 3.1) pain subscore (WOMAC Pain) at Week 12. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Pain subscore is standardized and reported ranging from 0 to 100 [0 = no pain, 100 = pain as bad as it can be].
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 103 | 98 | 100 | 101 | 101 | 106
score on a scale | -25.8 (20.5) | -29.3 (21.5) | -22.1 (20.2) | -32.1 (21.2) | -23.7 (24.6) | -22.8 (23.2)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.473, ANCOVA; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-7.99 to 3.72]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.040, ANCOVA; Mean Difference (Final Values) = -6.31, 95% CI 2-sided [-12.33 to -0.29]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.577, ANCOVA; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-4.35 to 7.79]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = -8.95, 95% CI 2-sided [-14.90 to -3.01]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.947, ANCOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-6.37 to 5.96]

7. Other Pre Specified Outcome: Change From Baseline OA Function in the Target Knee as Assessed by WOMAC Physical Function Subscore (WOMAC Function)
Description: Change from baseline OA function in the target knee as assessed by WOMAC Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function) at Week 12. The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore is standardized and reported ranging from 0 to 100 [0 = no functional disability, 100 = unable to function].
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 103 | 98 | 100 | 101 | 101 | 106
score on a scale | -26.0 (19.0) | -29.3 (21.8) | -20.9 (20.2) | -30.4 (21.3) | -22.7 (23.2) | -22.7 (24.2)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.299, ANCOVA; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-8.83 to 2.73]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = -7.18, 95% CI 2-sided [-13.24 to -1.12]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.675, ANCOVA; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-4.75 to 7.33]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Final Values) = -8.63, 95% CI 2-sided [-14.70 to -2.55]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.925, ANCOVA; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-5.99 to 6.59]

8. Other Pre Specified Outcome: Change From Baseline OA Pain in the Target Knee as Assesses by the Weekly Average of Daily Pain NRS
Description: Change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 12. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain (pain as bad as one can imagine).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 103 | 102 | 101 | 101 | 105 | 105
score on a scale | -2.75 (2.22) | -3.02 (2.03) | -2.21 (2.23) | -2.87 (2.10) | -2.15 (2.39) | -2.27 (2.27)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.062, ANCOVA; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.18 to 0.03]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.54 to -0.37]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.693, ANCOVA; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.75 to 0.50]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.39 to -0.17]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.697, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.49 to 0.74]

9. Other Pre Specified Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment (PtGA)
Description: Change from baseline OA disease activity as assessed by PtGA at Week 12. The PtGA completed using a 100 mm visual analog scale (VAS) adapted from the Patient Assessment Form © 1999, American College of Rheumatology. The subject rated how well he/she was doing, considering all the ways in which illness and health conditions may affected him/her. The VAS scale was anchored by "Very Well" on the left (scored as 0) and "Very Poorly" on the right (scored as 100). Higher scores indicated poorer disease assessment by the subject.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham
Number analyzed (Participants) | 100 | 93 | 94 | 101 | 99 | 104
score on a scale | -16.2 (25.0) | -20.0 (28.0) | -10.9 (23.4) | -18.4 (24.9) | -12.7 (21.9) | -12.7 (22.9)
Statistical Analysis 1: Comparison: 0.03 mg SM04690 vs Placebo; Test type: Superiority; p = 0.254, ANCOVA; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-9.04 to 2.40]
Statistical Analysis 2: Comparison: 0.07 mg SM04690 vs Placebo; Test type: Superiority; p = 0.031, ANCOVA; Mean Difference (Final Values) = -6.86, 95% CI 2-sided [-13.10 to -0.63]
Statistical Analysis 3: Comparison: 0.15 mg SM04690 vs Placebo; Test type: Superiority; p = 0.616, ANCOVA; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-7.20 to 4.28]
Statistical Analysis 4: Comparison: 0.23 mg SM04690 vs Placebo; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Final Values) = -7.62, 95% CI 2-sided [-13.41 to -1.82]
Statistical Analysis 5: Comparison: Placebo vs Sham; Test type: Superiority; p = 0.961, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-5.74 to 5.46]

ADVERSE EVENTS:
Time Frame: Data regarding treatment-emergent adverse events (TEAEs) was collected in this study. TEAEs are events that occur during the course of the study that are not present prior to Day 1 study medication injection, or, if present at the time of study medication injection, have worsened in severity during the course of the study. TEAEs were assessed at each study visit from the time of study medication injection on study visit Day 1 through Week 24 (End-of-Study)/Early Termination.
Description: The Safety Analyses Set [SAS] includes all subjects who received a study injection, analyzed as treated. Discrepancy in subject counts between SAS and Full Analysis Set [FAS] is the result of subjects who received a treatment that is different from the planned treatment group as randomized. Subjects who received a study treatment not as prescribed in the pharmacy manual are summarized in the "Other" treatment group for safety analysis reporting.
Groups:
- Other: Single intra-articular injection of an unidentified dose of SM04690 or Placebo due to incorrectly performed dilution or documentation by a pharmacist.
Arm/Group | 0.03 mg SM04690 | 0.07 mg SM04690 | 0.15 mg SM04690 | 0.23 mg SM04690 | Placebo | Sham | Other
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/104 | 0/106 | 0/106 | 0/114 | 0/120 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/106 | 0/104 | 0/106 | 2/106 | 1/114 | 0/120 | 1/39
Other Adverse Events (participants affected / at risk) | 14/106 | 19/104 | 14/106 | 17/106 | 15/114 | 22/120 | 9/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03 mg SM04690 (N=106) | 0.07 mg SM04690 (N=104) | 0.15 mg SM04690 (N=106) | 0.23 mg SM04690 (N=106) | Placebo (N=114) | Sham (N=120) | Other (N=39)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.03 mg SM04690 (N=106) | 0.07 mg SM04690 (N=104) | 0.15 mg SM04690 (N=106) | 0.23 mg SM04690 (N=106) | Placebo (N=114) | Sham (N=120) | Other (N=39)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 4 (4) | 4 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (8) | 2 (2) | 9 (12) | 3 (3) | 7 (7) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03122860/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03122860/SAP_001.pdf